CLINICAL TRIAL: NCT04121754
Title: Post-Stroke Walking Speed and Community Ambulation Conversion, A Pivotal Study
Brief Title: Post-Stroke Walking Speed and Community Ambulation Conversion Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedRhythms, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PS100
Record Dates: First submitted 2019-10-07; First posted 2019-10-10 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Chronic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Investigational Device (Experimental): Will walk for 30 minutes at a time, 3 times a week, for 5 weeks using the investigational device.
  Interventions: Device: MR-001
- Active Walking Control (Active Comparator): Will walk for 30 minutes at a time, 3 times a week, for 5 weeks using only foot sensors.
  Interventions: Other: Active Walking

INTERVENTIONS:
Device: MR-001 — Participants will walk using the investigational device (foot sensors, mobile device with mobile app and headphones) for thirty (30) minutes at a time, 3 times a week for 5 weeks.
  Other Names: Digital Rhythmic Auditory Stimulation Delivering Device
  Arms: Investigational Device
Other: Active Walking — Participants will walk for thirty (30) minutes at a time, 3 times a week for 5 weeks. No mobile devices, music players or headphones will be allowed. They will wear foot sensors during their active walking sessions to measure gait biomechanics.
  Arms: Active Walking Control

SUMMARY:
The purpose of this randomized, controlled study is to collect performance data on the ability of an investigational device designed to digitally deliver Rhythmic Auditory Stimulation to improve walking speed in people who suffered a stroke greater than six (6) months in the past and who are limited in mobility outside the home. The primary outcomes will be the mean change in walking speed (meters per second) and mean percent change in walking speed as determined by a 10-meter Walk Test after five weeks of intervention and compared between groups.

DETAILED DESCRIPTION:
Study participants who take part in this research study will participate in a screening visit, fifteen (15) intervention visits over approximately five weeks and a final closing visit. Study participants will be assigned by chance to one of the two study groups. Participants will not be able to switch groups once they are assigned. The investigational device includes a mobile device app and sensors that are attached to shoes. Headphones and a mobile device are also required to be used and will be provided in this study.

ELIGIBILITY:
Inclusion Criteria:

1. 50 years of age and older
2. Equal to or greater than six months post-stroke
3. A comfortable walking speed greater or equal to 0.5 meters per second (m/s), but less than 0.8m/s, as determined by a 10-meter walk test.
4. Demonstrates some level of asymmetry in gait

Exclusion Criteria:

1. Has a known history of neurologic (excluding stroke) injury
2. Has had more than 2 falls in the previous month
3. Is enrolled in another walking rehabilitation intervention (e.g., physical therapy)
4. Has an external lower limb prosthetic ("artificial limb")
5. Has a hearing impairment
6. Had orthopedic surgery in the last year
7. Has severe aphasia and/or a speech/language disorder
8. Has co-morbidities that prevent participation in exercise

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
Mean Change in Gait Speed measured by the 10-Meter Walk Test | Baseline through study completion, an average of six weeks
  Mean change in gait speed (meters per second) measured by the 10-Meter Walk Test compared between groups.
Mean Percent Change in Gait Speed measured by the 10-Meter Walk Test | Baseline through study completion, an average of six weeks
  Mean percent change in gait speed (meters per second) measured by the 10-Meter Walk Test compared between groups.

SECONDARY OUTCOMES:
Community Ambulation Status measured by the 10-Meter Walk Test | At study completion, an average of six weeks
  Gait speed (meters per second) measured by the 10-Meter Walk Test is equal to or greater than 0.8m/s.
Change in Cadence (steps per minute) as measured by a validated, instrumented walkway system | Baseline through study completion, an average of six weeks
  Cadence as measured by a validated, instrumented walkway system.
Change in Stride Length (meters) as measured by a validated, instrumented walkway system | Baseline through study completion, an average of six weeks
  Stride Length as measured by a validated, instrumented walkway system.
Change in Temporal Symmetry (percent) as measured by a validated, instrumented walkway system | Baseline through study completion, an average of six weeks
  Temporal Symmetry as measured by a validated, instrumented walkway system.
Change in Spatial Symmetry (percent) as measured by a validated, instrumented walkway system | Baseline through study completion, an average of six weeks
  Spatial Symmetry as measured by a validated, instrumented walkway system.
Change in Quality of Life as measured by the Stroke-Specific Quality of Life Scale (SS-QOL) | Baseline through study completion, an average of six weeks
  Change in quality of life as measured by the Stroke-Specific Quality of Life scale. Study participants must respond to each question of the SS-QOL with reference to the past week. It is a self-report scale containing 49 items in 12 domains and subscales which include: Energy, Upper extremity function, Work/Productivity, Mood, Self-care, Social roles, Family roles, Vision, Language, Thinking and Personality. Patients must respond to each item using the corresponding response set as indicated on 5 point scale. Higher scores indicate better functioning. The SS-QOL yields both domain scores and an overall SS-QOL summary score. The domain scores are unweighted averages of the associated items while the summary score is an unweighted average of all twelve domain scores.
Change in self-perceived disability as measured by the Stroke Impact Scale (SIS), Version 3.0 | Baseline through study completion, an average of six weeks
  Change in self-perceived disability as measured by the Stroke Impact Scale (SIS), Version 3.0. The scale includes 59 items and assesses 8 domains: Strength, Hand function, ADL/IADL, Mobility, Communication, Emotion, Memory and thinking, Participation/Role function. Each item is rated using a 5- point Likert scale in terms of the difficulty the patient has experienced in completing each item. It also includes the assessment of post-stroke recovery perception with a visual analog scale of 0-100 points (0: no improvement, 100: complete recovery).

CONTACTS AND LOCATIONS:
Overall Officials: Louis Awad, PT, DPT, PhD, Principal Investigator — Boston University
Locations (8):
- United States (8):
  - Shirley Ryan AbilityLab, Chicago, Illinois
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Trustees of Boston University, Boston, Massachusetts
  - Spaulding Rehabilitation Hospital, Charlestown, Massachusetts
  - Kessler Foundation, West Orange, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Atrium Health/Carolinas Rehabilitation, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No